CLINICAL TRIAL: NCT02733692
Title: Culturally Congruent HIV Risk Reduction App for Young Women, an Acceptability & Pilot Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 381039
Record Dates: First submitted 2016-01-11; First posted 2016-04-11 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: HIV; STDs
Keywords: HIV; STDs; web-based app; women
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Clinical Coding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GURHL Code Smartphone application (Experimental): Experimental arm will receive the 'Understanding Reproductive Health for Ladeez (GURHL) Code 'app' (application) for their smartphone with sexual health information. The intervention is embedded in the smart phone application. This includes sexual and reproductive health knowledge, plus access to a National Planned Parenthood health educator, and directions to other nearby clinics. Participants will be assessed using A-CASI at 3 months after enrollment.
  Interventions: Behavioral: Understanding Reproductive Health for Ladeez (GURHL) Code
- Control (No Intervention): The control arm will receive usual care. That is, they will receive a web-based flyer. This flyer will include a list of clinics and other trusted available resources, but without hyperlinks.
  Participants will be assessed using A-CASI at 3 months after enrollment.

INTERVENTIONS:
Behavioral: Understanding Reproductive Health for Ladeez (GURHL) Code — Understanding Reproductive Health for Ladeez (GURHL) Code is an acceptability study to test a web-based application designed with and for young women of color 18 to 25 years old.
  Arms: GURHL Code Smartphone application

SUMMARY:
Smartphone applications and mobile technologies offer users the potential to access critical information (e.g., proper condom use, directions to testing sites, and other sexual and reproductive health services) when it is needed most. Relevant findings will identify areas where existing interventions may be leveraged and adapted to work among young women of color in an urban setting and their networks. As SRH smartphone apps continue to proliferate, this study will expand researchers', developers', and health educators' limited knowledge about the feasibility, acceptability and preliminary efficacy of a sexual health educational app tailored with and for young Black and Latino women, aged 18-25 in NYC, including whether this app acts as a gateway to sexual health educators, clinical and other service providers. If proven effective, findings from this study will identify areas where existing interventions may be leveraged and adapted to work among a YBLW and their networks, and potentially adapted for other high needs communities.

DETAILED DESCRIPTION:
New HIV, Chlamydia and Gonorrhea infections are highest among young Black women and Latinas aged 13 to 29 years old compared to White women, which negatively impacts other sexual and reproductive health outcomes. Given that young women have a substantial need for SRH services and a high smartphone ownership, unique opportunities to utilize mobile apps(applications) to decrease HIV risk behaviors may exist.

A tailored, culturally congruent, smartphone app co-developed with and for young Black and Latino women (18 to 25 years old) not yet publicly available offers a unique opportunity to conduct a feasibility, acceptability, and pilot RCT. Using this app, this pilot that will: a) assess feasibility of the sampling, consent, recruitment and retention techniques; b) collect acceptability and usability data and cultural congruence on the app; a and c) collect pilot data to test differences between intervention and control groups on the preliminary estimates of app effectiveness to inform a potential larger-scale study. The investigators propose YBLW between 18 and 25 years old in NYC will use a mobile-based health education app to access SRH education information. Additionally, those who use the tailored SRH app will have more self-reported connection to SRH services, better knowledge of SRH education domains, and how to link to clinical services (e.g., PREP, PEP, EC, birth control, HIV, STD, and pregnancy testing), compared to the control group. Analysis for the first aim will employ process measures and the second and third aims are mixed-methods aims.

Analysis will compare differences between the 2-arms and indiscernible differences and culturally tailored usability will be explored via focus groups and web analytics.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 25 years old;
* self-identify as either Black and/or Latina;
* own a smartphone (iOS or android);
* live in NYC;
* report vaginal or anal intercourse in their lifetime;
* report unprotected intercourse in their lifetime;
* healthy (not controls) adults. There will be estimated total 110 of said subjects.

Exclusion Criteria:

* being married or partnered for more than one year,
* report only being sexually active with women,
* pregnant or have children 2 years old or younger,
* HIV+ status,
* men,
* individuals under 18 and over 25,
* live in a place other than New York City,
* formal training as a sexual peer health educator (beyond a high school health class) or
* unable to read English.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Preliminary Efficacy1 Improvement in Sexual Health Knowledge Condom Use | 3 months
  Effectiveness of the app based on reported knowledge of where to get condoms and how to use properly.
Preliminary Efficacy 2 Improvement in Sexual Health Knowledge Sexual and Reproductive Health Services | 3 months
  Effectiveness of the app based on reported knowledge of what sexual and reproductive health services exist and where to access them
Preliminary Efficacy 2 Improvement in Sexual Health Knowledge HIV and STD | 3 months
  Effectiveness of the app based on reported knowledge of what behaviors increase the risk for HIV and other sexually transmitted diseases
Preliminary Efficacy 3 Improvement in Sexual Health Knowledge Connection to Services | 3 months
  Effectiveness of the app based on reported knowledge of connection to sexual and reproductive health clinical services, based on whether women communicated with a reproductive health educator and whether she sought sexual and reproductive health services in person.

SECONDARY OUTCOMES:
Usability 1 Number of Times Used | 3 months
  The usability of the app will be determined by the number of times the app is opened
Usability 2 Actions Taken | 3 months
  The usability of the app will be determined by the actions users take during sessions (each action coded as positive regardless of which one, including other links clicked on, audio listened to or video links clicked on)
Usability 3 Duration | 3 months
  The usability of the app will be determined by the duration of page visits
Usability 4A App performance | 3 months
  The usability of the app will be determined by the number of technical errors encountered by users.
Usability 4B Ease of App usage | 3 months
  The usability of the app will be determined by the ease of usage and if users liked and understood the contents
Usability 5 Facilitators and Barriers | 3 months
  The usability of the app will be determined by user reports of facilitators and barriers to usage.
Usability 6 User Friendliness | 3 months
  The usability of the app will be determined by the users' assessment of usefulness, trustworthiness and usability

CONTACTS AND LOCATIONS:
Overall Officials: Denis Nash, PhD, Study Chair — CUNY Graduate School of Public Health & Health Policy
Locations (1):
- CUNY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The data collected and used ofr this will not be made publicly available.